CLINICAL TRIAL: NCT05202249
Title: Effect of Muscle and Skin Fixation of Thoracic Drainage Tube on Postoperative Pain in Patients Undergoing Uniport Thoracoscopic Pulmonary Resection
Brief Title: Effect of Muscle and Skin Fixation of Thoracic Drainage Tube on Postoperative Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Kun Li, MD, Kun Li, MD, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Kli4
Record Dates: First submitted 2022-01-09; First posted 2022-01-21 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Lung Neoplasms; Lung Cancer; Pulmonary Neoplasm; Postoperative Pain; Thoracoscopic Surgery
Keywords: chest tube drainage; thoracic drainage; thoracoscopic surgery; Postoperative Pain
MeSH Terms: conditions — Lung Neoplasms; Pain, Postoperative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- muscle layer fixation group (Experimental)
  Interventions: Procedure: muscle layer fixation of thoracic drainage tube
- conventional skin fixation group (No Intervention)

INTERVENTIONS:
Procedure: muscle layer fixation of thoracic drainage tube — The thoracic drainage tube is fixed on the muscle layer of the uniport
  Arms: muscle layer fixation group

SUMMARY:
Lung cancer is the leading cause of cancer-related death worldwide. Thoracoscopic pulmonary resection is a prevalent management for early stage of lung cancer. Placement of chest tube is the standard procedure after surgery, which causes pain that cannot be ignored. The investigators aimed to determine whether a muscle layer fixation of thoracic drainage tube could release postoperative pain in patients with uniport thoracoscopic pulmonary resection compared with conventional skin fixation.

ELIGIBILITY:
Inclusion Criteria:

* 18<age<80;
* ASA≤III
* Patients with no clinically significant cardiac history, such as ischaemic heart disease, valvular heart disease, rhythm disturbances such as frequent atrial fibrillation or premature ventricular contractions (PVCs). Patients with significant cardiac history should be optimized according the relevant guidelines before surgery is considered.
* Normal cardiopulmonary function [predicted forced expiratory volume in the first second(FEV1%) >50% and ejection fraction (EF) >50%of predicted value]. Resting blood gas analysis showing arterial partial pressure of oxygen (PaO2)≥75 mmHg and arterial partial pressure of carbon dioxide (PaCO2) <45 mmHg;

Exclusion Criteria:

* History of ipsilateral surgery and other conditions which can result in extensive pleural adhesion;
* Coagulopathy, hypoxemia (PaO2 <60 mmHg), hypercapnia [arterial carbon dioxide tension(PaCO2) >50 mmHg];
* Significant cardiac history.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-03-15 (Estimated); Study Completion 2022-05-15 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain | From date of operation until the date of chest tube removal, assessed up to 7 days
  The postoperative pain is assessed using a Visual Analog Scale (VAS)
Pain-associated inflammatory factor | the first day after surgery
  the level of pain-associated inflammatory factor in blood, including CRP, PCT, IL6 and TNFa
Dosage of analgesics | From date of operation until the date of chest tube removal, assessed up to 7 days
  Dosage of analgesics

CONTACTS AND LOCATIONS:
Locations (1):
- Daping Hospital and the Research Institute of Surgery of the Third Military Medical University, Chongqing, Chongqing Municipality, China